CLINICAL TRIAL: NCT02315339
Title: European Home Mechanical Ventilation Registry
Acronym: EHMVR
Status: Terminated | Type: Observational
Sponsor: ResMed (Industry)
Collaborators: Clinical Trial Center North Hamburg Germany (Unknown); CRI-The Clinical Research Institute GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: CTC11633
Record Dates: First submitted 2014-10-06; First posted 2014-12-11 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Amyotrophic Lateral Sclerosis; Spinal Cord Injury; Muscular Dystrophies; Obesity Hypoventilation Syndrome; Kyphoscoliosis; Congenital Central Hypoventilation Syndrome; Duchenne Muscular Dystrophy; Myopathies; Myotonic Dystrophy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Muscular Dystrophies; Obesity Hypoventilation Syndrome; Congenital central hypoventilation syndrome; Muscular Dystrophy, Duchenne; Muscular Diseases; Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The European Home Mechanical Ventilation Registry (EHMVR) will enable a thorough evaluation of HMV by documenting the characteristics of HMV patients and their treatment. This will facilitate a prospective, observational study to identify the primary indications for HMV, describe patterns of HMV use in European countries, and characterize changes in the initiation and utilization of HMV over time. The registry will target all adult individuals who have an indication for HMV. In the EHMVR, patient data from routine clinical care will be documented using an electronic case report form (eCRF). The eCRF will record: patient demographic data; diagnostic information (including primary diagnosis, 6-minute walk time, the presence of depression, and quality of life); blood gases; ventilation treatment (including type of ventilator, modes and settings, interfaces used); follow-up data (including failure rates, side effects, technical issues). An initial Pilot Phase will be launched with the aim to enrol at least 200 patients over a 6-month period to determine the feasibility of the registry. Steering committee members and their institutions will be the main participants in the Pilot Phase. After completion of the Pilot Phase, the registry will be expanded across Europe with the goal of enrolling approximately 10,000 patients over 5 years.

DETAILED DESCRIPTION:
The data (baseline and follow-up) should be collected as part of routine clinical care. In clinical practice, after HMV initiation, the first control examination (follow-up number one) with nocturnal diagnostics should take place within the first 4-8 weeks. Annual follow-up is required, and it is recommended that subsequent control visits should be performed 1-2 times a year. Each patient will be included for 5 years (total duration of the registry).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with an indication to receive HMV as part of routine clinical care
* Patient is able to fully understand the study information and is willing to give informed consent
* Patient, or the patient's legal guardian, signing the consent form

Exclusion Criteria:

- No exclusion criteria have been defined because only data from routine clinical care are needed, plus a separate healthcare questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry will target all adult individuals who have an indication for HMV (including those with amyotrophic lateral sclerosis [ALS], central hypoventilation syndrome [CHS], chronic obstructive pulmonary disease [COPD], kyphoscoliosis, obesity hypoventilation syndrome [OHS], spinal cord injury [SCI], Duchenne muscular dystrophy [DMD], muscular dystrophies [MDs] other than DMD, myopathies and myotonic dystrophy [Steinert's muscular dystrophy; SMD]). All newly-diagnosed patients with chronic respiratory diseases who are eligible for HMV treatment as part of routine care can be included in the registry. Patients who satisfy all the inclusion criteria will be consecutively enrolled into the registry.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Determine the mortality rate and the number of hospital readmissions | every year (2014 to 2019), up to 5 years

SECONDARY OUTCOMES:
Determine the effects of home mechanical ventilation on health-related quality of life using the EQ-5D and the Severe Respiratory Insufficiency questionnaires quality of life | every year (2014 to 2019), up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pepin, Pr, Principal Investigator — Laboratoire d'EFCR, RDC Haut Chartreuse, CHU Michallon 38043,Grenoble, France; Stefano Nava, Pr, Principal Investigator — Pneumologia e Terapia Intensiva Respiratoria Ospedale Sant' Orsola Malpighi, Italy; Anita Simonds, Pr, Principal Investigator — NIHR Respiratory Biomedical Research Unit, Royal Brompton and Harefield NHS Foundation Trust, United Kingdom; Wolfram Windisch, Pr, Principal Investigator — Lungen Klinik - Chefarzt Abt. Pneumologie Kliniken der StadtKölng GmbH, Ostmerheimer Strasse 200, Germany
Locations (1):
- Lungen Klinik - Chefarzt Abt. Pneumologie Kliniken der StadtKölng GmbH, Cologne, Germany